CLINICAL TRIAL: NCT01601951
Title: Autologous Bone Marrow Concentrate Database Outcomes Research Project
Brief Title: Outcomes Data of Bone Marrow Stem Cells to Treat Hip and Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Regenerative Pain Center, Illinois (Other)
Responsible Party: Sponsor
Other Study IDs: MM-01
Record Dates: First submitted 2012-05-14; First posted 2012-05-18 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Hip and Knee Osteoarthritis
Keywords: Osteoarthritis; Stem Cell Injections; Bone Marrow; Autologous
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hip Osteoarthritis
  Interventions: Other: Procedural, Bone Marrow concentrate injection
- Knee Osteoarthritis
  Interventions: Other: Procedural, Bone Marrow concentrate injection

INTERVENTIONS:
Other: Procedural, Bone Marrow concentrate injection — This is strictly data collection and outcomes based. The procedure is not part of this study

SUMMARY:
The purpose of this study is to determine if Bone Marrow Concentrate may be successful in the treatment of osteoarthritis. Bone Marrow Concentrate is known to contain a community of cells that has been shown to have "regenerative" properties. This study is designed to evaluate the short-term clinical and x-ray outcomes of injections for hip and knee osteoarthritis.

Inclusion Criteria:

* Subjects must be scheduled for an autologous bone marrow hip or knee injection
* Subjects must have a diagnosis of hip or knee osteoarthritis
* Subjects must be between the ages of 18 and 85
* Subjects must be willing and able to sign Informed Consent
* Subjects must be willing and able to return for scheduled follow-up evaluations

Exclusion Criteria:

* Subjects who have had any type of visco-supplementation in the treated joint within the last three months prior to enrollment
* Subjects for whom baseline data is not available

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be scheduled for an autologous bone marrow hip or knee injection
* Subjects must have a diagnosis of hip or knee osteoarthritis
* Subjects must be between the ages of 18 and 85
* Subjects must be willing and able to sign Informed Consent
* Subjects must be willing and able to return for scheduled follow-up evaluations

Exclusion Criteria:

* Subjects who have had any type of visco-supplementation in the treated joint within the last three months prior to enrollment
* Subjects for whom baseline data is not available

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Orthopedic clinic, those with a diagnosis of hip or knee osteoarthritis, scheduled for an Autologous Bone Marrow injection
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2012-04; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Visual Analog Pain Scale | Baseline, 6 weeks, 3 months, 1 year
  Change in subjective pain measure
Harris Hip Score or Knee Society Score | Baeline, 6 weeks, 3 months, 1 year
  Change in subjective pain, function, functional activity measurement and a clinical physical exam
Physician Global Assessment | Baseline, 6 weeks, 3 months, 1 year
  Change in physician rated disease activity measurement

SECONDARY OUTCOMES:
Radiologic | Baseline, 1 year
  Radiographic changes of the hip or knee

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Sheinkop, M.D., Principal Investigator — Regenerative Pain Center
Locations (1):
- Regenerative Pain Center, Des Plaines, Illinois, United States